CLINICAL TRIAL: NCT03869463
Title: Testing the Mechanism of Action of Computerized Cognitive Training in Young Adults With Depression: Clinical, Cognitive and Neuroimaging Outcomes
Brief Title: Computerized Cognitive Training in Young Adults With Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Challenges to recruitment
Sponsor: Queens College, The City University of New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2018-1311
Record Dates: First submitted 2019-02-07; First posted 2019-03-11 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2022-09

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EF/PS CCT (Experimental): This group will complete EF/PS (executive functioning/processing speed) computerized cognitive training (CCT) which includes games specifically focused on executive function & processing speed.
  Interventions: Other: Computerized Cognitive Training
- Verbal CCT (Active Comparator): This group will complete verbal-focused computerized cognitive training.
  Interventions: Other: Computerized Cognitive Training
- Waitlist Control (Placebo Comparator): This group will not receive cognitive training during study participation.
  Interventions: Other: Control

INTERVENTIONS:
Other: Computerized Cognitive Training — Participants will complete 8 weeks of computerized cognitive training through the Peak platform on mobile devices.
  Arms: EF/PS CCT; Verbal CCT
Other: Control — This group will not receive computerized cognitive training.
  Arms: Waitlist Control

SUMMARY:
The purpose of the study is to examine the benefits and mechanism of action of computerized cognitive training (CCT) on mood, neuropsychological deficits, everyday functioning, and brain activity among young adults with a range of depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-29.
2. Current diagnosis of MDD/persistent depressive disorder or HDRS greater than or equal to 12. 3. Daily access to smartphone or tablet with internet connection for the study duration.

4. Willing and able to complete MRI, mood, and neuropsychological testing. 5. IQ > 85.

Exclusion Criteria:

1. Lacks English-speaking ability as determined by self-report and clinical evaluation.
2. Evidence of schizophrenia, schizoaffective disorder, psychosis, bipolar I and II disorder.
3. Active suicidal ideation, intent, or plan, or past attempt within 1 year.
4. Severe depression (HDRS > 30).
5. Neurological disorder (epilepsy, multiple sclerosis, traumatic brain injury, clinical stroke).
6. Use of medications known to have negative impact on cognition (benzodiazepines and lorazepam equivalents > 1mg daily, narcotics, anticholinergics).
7. History of alcohol or drug abuse or dependence within past year.
8. Acute, severe, unstable medical illness. For cancer, acutely ill patients (including those with metastases) are excluded, but past history of successfully treated cancer does not result in exclusion.
9. Regular online brain training or regular player of non-fluency verbal games, defined as doing these procedures at a frequency of twice weekly or greater during the year prior to screening.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Sheehan Disability Scale | Screen, Week 0, Week 4, Week 8, 3-month follow-up
  Self-report questionnaire of everyday functioning. It includes three subscales: work, social life, leisure activities, and home life or family responsibilities. Each subscale is rated on a 10-point scale for a minimum total score of 0 and a maximum total summed score of 30 across the three subscales. High scores are associated with more impairment.
Change in Hamilton Depression Rating Scale | Screen, Week 0, Week 4, Week 8, 3-month follow-up
  Clinician-rated measure of depression composed of 21 questions. The first 17 items are scored: eight items have a 5-point scale, nine items have a 3-point scale. Total score range is 0-52. Higher scores indicate more severe symptoms.
Change in DKEFS Trail Making Test - Condition 4 | Weeks 0, 4, 8, 3-month follow- up
  Measure of executive function. It is a switching task that requires the subject to connect numbers and letters in an alternating pattern (1-A-2-B, etc.) as quickly as possible.
Change in Emotional Go/No Go Task (fMRI) | Week 0, Week 4 or Week 8 (depending on randomization)
  Measure of behavioral inhibition and set shifting. Participants must press a button for pre-specified to go trials and withhold pressing the button for pre-specified no-go trials.

SECONDARY OUTCOMES:
Change in Beck Depression Inventory-II | Screen, weekly for weeks 0-8, 3-month follow-up
  Self-report questionnaire of depression composed of 21 questions on a 4-point scale. Total score ranges from 0-63. Higher scores indicate worse symptom severity.
Change in WAIS-IV Coding | Weeks 0, 4, 8, 3-month follow- up
  Participants are required to copy symbols paired with numbers in a 120 second time limit. The score is the number correct in the allotted time.
Change in Connectivity Index (resting state fMRI) | Week 0, Week 4 or Week 8 (depending on randomization)
  Measure of resting state fMRI. Higher scores indicate more connectivity within the network

OTHER OUTCOMES:
Change in DKEFS Trail Making Test - Condition 2 | Weeks 0, 4, 8, 3-month follow- up
  Measure of processing speed. This is a paper and pencil test requiring subjects to connect in order 25 encircled numbers randomly arranged using pencil lines.
Change in DKEFS Color-Word Interference Test | Weeks 0, 4, 8, 3-month follow- up
  Measure of response inhibition. This test is divided into four sections: color naming, word reading, color-word inhibition, and color-word inhibition/ switching. The score in each condition is the completion time as well as the number of errors and self-corrections.
Change in WAIS-IV Digit Span Forwards | Weeks 0, 4, 8, 3-month follow- up
  Measure of attention. This test requires participants to repeat back strings of digits in the same order in which they heard them.
Change in WAIS-IV Digit Span Backwards | Weeks 0, 4, 8, 3-month follow- up
  Measure of working memory. This test requires participants to repeat back strings of digits in the reverse order in which they heard them.
Change in WAIS-IV Symbol Search | Weeks 0, 4, 8, 3-month follow- up
  Measure of processing speed. Subjects are required to visually scan and mark off the same object as a target stimulus among a set of distractors in a 120 second time limit.
Change in DKEFS Letter and Category Naming Test | Weeks 0, 4, 8, 3-month follow- up
  Measure of verbal fluency. This test requires subjects to generate words that begin with a particular letter or belong to a particular semantic category as quickly as possible. Total score is the number of words generated in 60 seconds per trial.
Change in California Verbal Learning Test-II | Weeks 0, 4, 8, 3-month follow- up
  Measure of short-term and long-term verbal memory. For this test, the participant is read a list of words five times. He/she is asked to recall what was on the list immediately after each reading of the list. After a delay, the participant is again asked to recall what words were on the list.
Change in Brief Visuospatial Memory Test-Revised | Weeks 0, 4, 8, 3-month follow- up
  Measure of visual spatial memory. Subjects reproduce a series of six designs on paper, visually presented for 10 seconds on three trials. After a delay, the subject is asked to recall the presented designs again.

CONTACTS AND LOCATIONS:
Overall Officials: Joel R Sneed, PhD, Principal Investigator — Professor
Locations (1):
- Queens College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rushia SN, Schiff S, Egglefield DA, Motter JN, Grinberg A, Saldana DG, Shehab AAS, Fan J, Sneed JR. Testing the Mechanism of Action of Computerized Cognitive Training in Young Adults with Depression: Protocol for a Blinded, Randomized, Controlled Treatment Trial. J Psychiatr Brain Sci. 2020;5:e200014. doi: 10.20900/jpbs.20200014. Epub 2020 Jun 19. PMID 32743079